CLINICAL TRIAL: NCT00126490
Title: Phase 2 Trial of Sequential Bevacizumab Then Subcutaneous Interleukin-2 in Metastatic Renal Cancer
Brief Title: Bevacizumab and Interleukin-2 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02663; NCI-2012-02663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000434852; NCI-6438; MCC-IRB-102782; MCC 13921 (Other: Moffitt Cancer Center); 6438 (Other: CTEP); P30CA076292 (NIH)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — aldesleukin; Bevacizumab; Immunoglobulin G; Disulfides

ARMS (1):
- Treatment (bevacizumab, aldesleukin) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 in weeks 1, 3, 5, 7, 9, and 11. Patients also receive interleukin-2 subcutaneously on days 1-5 in weeks 5-10. Treatment repeats every 12 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease then receive bevacizumab alone in weeks 1, 3, 5, 7, 9, and 11. Courses with bevacizumab alone repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Biological: Bevacizumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Aldesleukin — Given subcutaneously
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with interleukin-2 works in treating patients with metastatic kidney cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Interleukin-2 may stimulate the white blood cells to kill tumor cells. Giving bevacizumab together with interleukin-2 may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the frequency of major response in patients with metastatic renal cell cancer treated with bevacizumab and interleukin-2.

SECONDARY OBJECTIVES I. Compare the median progression-free survival and median overall survival of patients treated with this regimen with risk-stratified historical controls from published risk models.

OUTLINE:

Patients receive bevacizumab IV over 30-90 minutes on day 1 in weeks 1, 3, 5, 7, 9, and 11. Patients also receive interleukin-2 subcutaneously on days 1-5 in weeks 5-10. Treatment repeats every 12 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease then receive bevacizumab alone in weeks 1, 3, 5, 7, 9, and 11. Courses with bevacizumab alone repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days and then every 3 months for at least 2 years.

PROJECTED ACCRUAL: Approximately 10-38 patients will be accrued for this study within 21 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell cancer

  * Metastatic disease
  * More than 75% clear cell histology
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No prior refractory disease, defined as clinical or radiologic progression, during or within 3 months after completion of prior interleukin-2 (IL-2)
* Nominally "good" or "intermediate" risk disease, meeting ≥ 4 out of 5 of the following criteria:

  * Hemoglobin > 10 g/dL (except for patients with hereditary hemoglobinopathy)
  * ECOG performance status 0-1 (required)
  * Calcium normal (corrected)

    * Patients with hypercalcemia due to malignancy allowed provided it has been controlled for > 1 month
  * Primary tumor treated or resected by complete nephrectomy, partial nephrectomy, radiofrequency ablation, or other local ablation
  * Lactic dehydrogenase < 1.5 times upper limit of normal (ULN)
* No history of or current brain or CNS metastasis by CT scan or MRI within the past 30 days
* Performance status - ECOG 0-1
* More than 4 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* No history of bleeding diathesis
* PTT < 1.5 times ULN
* INR < 1.5
* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* No chronic hepatitis B or C
* Creatinine ≤ 2.0 mg/dL
* No proteinuria* by dipstick urinalysis
* Urine protein ≤ 1,000 mg by 24-hour urine collection
* No symptomatic congestive heart failure
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 160 mm Hg and diastolic BP > 90 mm Hg
* No cardiac arrhythmia
* No peripheral vascular disease ≥ grade 2
* No clinically significant peripheral artery disease
* None of the following arterial thromboembolic events within the past 6 months:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina pectoris
  * Myocardial infarction
* Not pregnant
* No nursing during and for 3 months after completion of study treatment
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for 3 months after completion of study treatment
* No active infection requiring parenteral antibiotics
* No known HIV positivity
* No history of allergic reaction to antibody drugs or IL-2
* No psychiatric illness or social situation that would preclude study compliance
* No non-healing wound or fracture
* No insulin-dependent diabetes
* No other uncontrolled illness
* No other malignancy requiring active treatment within the past 2 years except nonmelanoma skin cancer
* No prior bevacizumab
* At least 6 months since prior immunotherapy containing IL-2
* At least 2 months since prior investigational antibodies
* More than 4 weeks since prior conventional cytotoxic chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No concurrent corticosteroids except replacement corticosteroids for adrenal insufficiency OR inhaled steroids for chronic obstructive pulmonary disease, asthma, or allergic rhinitis
* More than 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to the only site of measurable disease unless there has been subsequent disease progression
* More than 4 weeks since prior major surgery
* At least 24 hours since prior minor surgical procedure, placement of vascular access device, or fine needle aspiration
* At least 30 days since prior and no other concurrent investigational agents
* More than 10 days since prior anticoagulants

  * Low-dose anticoagulants for maintenance of vascular access device patency allowed
* No concurrent therapeutic warfarin, including warfarin for treatment of deep vein thrombosis or pulmonary embolism
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-03; Primary Completion 2012-06 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayer Fishman, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began 03/23/2005 and accrual was closed 8/21/2007 due to slow accrual.
Pre-assignment Details: 24 enrolled but 5 were never treated (moved away, creatinine too high, Hospice before starting, lived too far away to come, chromophobe subtype after review of pathology)
Period: Overall Study
Arm/Group | Treatment (Bevacizumab, Aldesleukin)
Started | 19
Completed | 18
Not Completed | 1
Not completed — Stopped after 1 infusion (fall/injury) | 1

BASELINE CHARACTERISTICS:
Population: 18 of the 19 who started treatment were evaluable. One participant had to withdraw after only one infusion because they fell and broke both wrists.
Arm/Group | Treatment (Bevacizumab, Aldesleukin)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 66 [41 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Evaluable Participants With Complete Response (CR) and Partial Response (PR) at One Year
Description: Major response according to Response Evaluation Criteria In Solid Tumors (RECIST). CR: Disappearance of all target lesions; Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 1 year
Population: All Participants who received at least one treatment
Measure: Number; unit: participants
Groups:
- Treatment (Bevacizumab, Aldesleukin): Patients received bevacizumab IV over 30-90 minutes on day 1 in weeks 1, 3, 5, 7, 9, and 11. Patients also received interleukin-2 subcutaneously on days 1-5 in weeks 5-10. Treatment repeated every 12 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease then received bevacizumab alone in weeks 1, 3, 5, 7, 9, and 11. Courses with bevacizumab alone repeated every 12 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Bevacizumab, Aldesleukin)
Number analyzed (Participants) | 19
participants
  Complete Response | 0 [0 to 0]
  Partial Response | 1 [0.1 to 26.0]

2. Secondary Outcome: Number of Evaluable Participants With Overall Survival (OS) at 2 Years
Description: Overall Survival tabulation at 2 years from start of treatment.
Time Frame: 2 years from start of treatment
Population: Evaluable participants
Measure: Number; unit: participants
Arm/Group | Treatment (Bevacizumab, Aldesleukin)
Number analyzed (Participants) | 18
participants | 10

3. Secondary Outcome: Number of Evaluable Participants With Progression Free Survival (PFS)
Description: Progression Free Survival tabulation at 1 year and at 2 years. Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 2 years
Population: Evaluable participants
Measure: Number; unit: participants
Arm/Group | Treatment (Bevacizumab, Aldesleukin)
Number analyzed (Participants) | 18
participants
  PFS at 1 year | 3
  PFS at 2 years | 1

4. Secondary Outcome: Pearson Correlation Coefficients of Dendritic Cell (DC):Immature Cell (ImC) Ratio With DC Function
Description: Dendritic cell (DC) phenotype or functionality. Pearson correlation coefficients of DC:ImC ratio with DC function were to be computed and tested for departure from zero. Those with major responses were to be compared to those without major responses with respect to baseline DC:ImC ratio, baseline DC functional assay, post-treatment DC:ImC ratio and post-treatment DC functional assay using pooled t tests.
Time Frame: At baseline, at days 4-5, 9-10 (of course 1), and at the end of treatment
Population: This was not evaluable because there were not enough samples.
Arm/Group | Treatment (Bevacizumab, Aldesleukin)
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Possibly Related Serious Adverse Events (SAEs)
Description: Number of Participants with Serious Adverse Events (SAEs) Possibly Related to Study Treatment. Toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Time Frame: Up to 30 days after completion of treatment
Population: All Participants who received at least one treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Bevacizumab, Aldesleukin)
Number analyzed (Participants) | 19
participants | 4

ADVERSE EVENTS:
Time Frame: 2 years
Description: "0" had to be entered for Other (not including Serious) Adverse Events, because they were not tabulated for treatment 3/30/05 through 1/24/07.
Arm/Group | Treatment (Bevacizumab, Aldesleukin)
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab, Aldesleukin) (N=19)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Death not associated with CTCAE term (General disorders) | 2 (2)
Thyroid function low, (hypothyroidism) (Endocrine disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Ulcer, GI - Stomach (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bone (osteomyelitis) (Infections and infestations) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) - Trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Pain - Joint (General disorders) | 1 (1)
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Investigators planned to have 38 participants treated on this study. "0" had to be entered for Other (not including Serious) Adverse Events, because they were not tabulated for treatment 3/30/05 through 1/24/07.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less